CLINICAL TRIAL: NCT02776306
Title: Effects of Mirror Box Therapy on Neuroplasticity and Functional Outcome in Hemiparetic Upper Limb Post Stroke
Brief Title: Mirror Box Imaging Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Collaborators: Anglia Ruskin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P0868
Record Dates: First submitted 2016-04-07; First posted 2016-05-18 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mirror box therapy (Experimental): The participants in the mirror box therapy arm will receive mirror box therapy for 3 weeks for upper limb rehabilitation post stroke.
  Interventions: Other: Mirror Box therapy
- Standard treatment group (No Intervention): The participants will receive the standard treatment arm for 3 weeks for upper limb rehabilitation post stroke.

INTERVENTIONS:
Other: Mirror Box therapy — In mirror box therapy the patient uses the reflection of their good arm to trick to brain into thinking that the effected arm is working.
  Arms: Mirror box therapy

SUMMARY:
The purpose of this study is to evaluate the effects of mirror box therapy on upper extremity, motor recovery and motor functioning in patients that have suffered a stroke.

DETAILED DESCRIPTION:
Arm and hand weakness as a result of stroke occurs in approximately 70% of stroke survivors, with 30%-60% of patients being unable to fully recover functional use of their upper limbs. As recovery may be due to insufficient or inadequate therapeutic interventions, the progress and evaluation of upper limb treatment is currently being investigated.

Mirror Box therapy is a task orientated, non-invasive, economic and patient directed therapy for hemiparetic upper limb post stroke patients. The study is intended to evaluate cerebral reorganization by using mirror therapy. Movements of the stronger limb trick the brain into thinking that the weaker arm is moving and to stimulate the respective brain areas.

Patients are enrolled into two groups using standard upper limb rehabilitation for three weeks followed by standard rehabilitation plus Mirror Box for another three weeks (Group 1). Group 2 will receive the same therapy in inverted order.

Patients will receive clinical and functional assessment at baseline, three weeks and six weeks including brain MRI using functional resting state MRI.

The primary outcome is functional connectivity (correlation coefficient) at baseline and after treatment. Secondary endpoints include motor and functional recovery using outcome measures like Fugl Meyer assessment, Action Research Arm Test, grip and pincer strength. Further secondary endpoints are increase in sensorimotor cortex activation across the period of therapy and cortical reorganization.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs to 105yrs
* Hemiparetic upper limb post stroke
* Capable of providing informed consent
* Intact vision: if diagnosis of peripheral field defect, patient should be able to compensate for it.

Exclusion Criteria:

* Any contraindication to MRI scanning
* Clinically significant psychiatric disorder (e.g. depression)
* Pre-existing neurological or psychiatric disease that could confound the study results.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Change in brain connectivity will be assessed by resting-state fMRI | Baseline, 3 weeks and at 6 weeks

SECONDARY OUTCOMES:
Activity of daily living will be assessed with Barthel index. | Baseline, 3 weeks and at 6 weeks
Function of the affected hemiplegic upper limb will be assessed with action research arm test | Baseline, 3 weeks and at 6 weeks
Impairment in the hemiplegic upper limb will be assessed with Fugl Meyer test. | Baseline, 3 weeks and at 6 weeks
Grip strength will be assessed using hand dynamometer | Baseline, 3 weeks and at 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iris Grunwald, Principal Investigator — Anglia Ruskin University
Locations (1):
- Southend Hospital, Westcliff-on-Sea, Essex, United Kingdom

IPD SHARING:
Plan to Share IPD: No